CLINICAL TRIAL: NCT00706498
Title: A Single Arm Phase II Study to Investigate the Efficacy, Safety and Pharmacokinetics of a Single Dose of 200 mg of i.v. BI 2536, Administered Once Every 3 Weeks in Patients With Advanced Metastatic Hormone-refractory Prostate Cancer.
Brief Title: Phase II Study of BI 2536 in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 1216.19
Record Dates: First submitted 2008-06-24; First posted 2008-06-27 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BI 2536

INTERVENTIONS:
Drug: BI 2536

SUMMARY:
A study to investigate the activity of BI 2536 in Prostate Cancer

ELIGIBILITY:
Inclusion Criteria:

* Male patient age >18 years.
* Signed informed consent.
* Able to comply with protocol requirements.
* Patients with histologically, cytologically or biochemically documented metastatic adenocarcinoma of the prostate, clinically refractory or resistant to hormone therapy, as documented by progression following at least one hormonal therapy, which must include orchidectomy or gonadotropin releasing hormone agonist (GnRHa).
* Patients with Progressive Disease (PD). PD is defined as a minimum of three consecutive serum PSA measurements obtained at least 7 days apart within the previous 3 months of start of trial, which document progressively increasing PSA values. Patients with progression of measurable disease (RECIST) or progression of bone disease must also fit the criterion for PSA progression.
* Patients must have documented progression (as defined above) following anti-androgen withdrawal of 4 weeks duration for flutamide and 6 weeks for bicalutamide or nilutamide. For a patient who has withdrawn from anti-androgen therapy less than 6 months prior to inclusion in the trial, one of the following criteria is also required:
* Following completion of the anti-androgen withdrawal period one PSA measurement should be higher than the last pre-withdrawal PSA.

Or

* Following the completion of the anti-androgen withdrawal period if the PSA value has decreased, a patient can still qualify if 2 increases in PSA are documented after the post- withdrawal nadir.
* PSA > 10 ng/ml.
* A predicted life expectancy of at least 12 weeks.
* A maximum of one prior treatment with either chemotherapy or other non-hormonal treatment modality.
* ECOG performance status 0-1.
* Stable analgesia requirements.
* INR Prothrombin time (PT) and partial thromboplastin time (PTT) <1.5 upper limit of normal.
* Adequate bone marrow function defined as absolute neutrophil count (ANC) > 1.5 x 109l, Platelet count > 100 x 109/l.
* Haemoglobin > 9.0 mg/dl.
* Serum Albumin > 2.0 g/l.
* Castrate testosterone level [< 20 ng/dl or <0.69nM (nM/L x 28.8 = ng/dl)] must be maintained during the duration of the trial by orchidectomy or medical castration.
* Patients on oral or intravenous bisphosphonates are allowed to enter the trial as long as they have been on bisphosphonates for a minimum of 3 months.

Exclusion Criteria:

* Prior treatment with more than one cytotoxic chemotherapy regimen.
* Known or suspected hypersensitivity to the trial drug or their excipients.
* Persistence of toxicities of prior anti-cancer therapies which are deemed to be clinically relevant.
* Aspartate amino transferase (ast) or alanine amino transferase (alt) greater than 2.5 times the upper limit of normal, or aspartate amino transferase (ast) or alanine amino transferase (alt) greater than 5 times the upper limit of normal in case of known liver metastases.
* Bilirubin greater than 1.5 mg/dl (> 26 micromol/l, Si unit equivalent). Serum creatinine greater than 2.0 g/l.
* Concomitant intercurrent illnesses including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situation that would limit compliance with trial requirement or which are considered relevant for the evaluation of the efficacy or safety of the trial drug.
* Systemic corticosteroids taken within the past 28 days before screening (inhaled corticosteroids prescribed for bronchospasm are allowed). Patients on long-term stable-dose steroids for concurrent illness are not excluded.
* Treatment with any investigational drug within 28 days of trial onset.
* History of other malignancies which could affect compliance with the protocol or interpretation of results within 5-years. Patients with adequately treated basal or squamous cell skin cancer are generally eligible.
* Patient with history or clinical evidence of CNS disease or brain metastases.
* Patients with symptoms of impending or established spinal cord compression.
* Radiotherapy within the past four weeks prior to treatment with the trial drug.
* Prior radioisotope therapy (except radium-223 which is permissible).
* Immunotherapy within the past four weeks prior to treatment with the trial drug.
* Patients unable to comply with the protocol.
* Active alcohol or drug abuse.
* Patients who do not use adequate contraception.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
PSA response rate at 12 weeks according to Prostate Specific Antigen Working Group (PSAWG) criteria. | 12 weeks

SECONDARY OUTCOMES:
PSA response duration | at least 12 weeks
Time to PSA progression assessed at 24 weeks | 24 weeks
Overall objective response using RECIST criteria (complete response [CR] or partial response [PR]) in patients with measurable disease | at least 12 weeks
Time to death | at least 12 weeks
Time to overall progression | at least 12 weeks
Progression free survival | at least 12 weeks
Overall survival | at least 12 weeks
Duration of overall response (RECIST) | at least 12 weeks
BI 2536 plasma concentrations | 1 week
Incidence and intensity of AEs, with grading according to the US National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, version 3.0) | 24 weeks
Number of patients with changes in laboratory safety parameters | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- United Kingdom (6):
  - 1216.19.4407 Boehringer Ingelheim Investigational Site, Cambridge
  - 1216.19.4405 Boehringer Ingelheim Investigational Site, Guildford
  - 1216.19.4402 Boehringer Ingelheim Investigational Site, Headington
  - 1216.19.4406 The Christie NHS Foundation Trust, Manchester
  - 1216.19.4404 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1216.19.4401 Boehringer Ingelheim Investigational Site, Sutton